CLINICAL TRIAL: NCT04998760
Title: A Multi-center Clinical Study to Evaluate Dual mTORC1/2 Inhibitor (ATG 008) or Selective Inhibitor of Nuclear Export Compound (ATG-010) in Combination With Chemotherapy in Patients With Relapsed or Metastatic Ovarian Cancer, Endometrial Cancer, and Cervical Cancer
Brief Title: A Study to Evaluate Dual mTORC1/2 Inhibitor (ATG 008) or Selective Inhibitor of Nuclear Export Compound (ATG-010) in Combination With Chemotherapy in Patients With Relapsed or Metastatic Ovarian Cancer, Endometrial Cancer, and Cervical Cancer ( PORCH )
Acronym: PORCH
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Qi Zhou (Other)
Responsible Party: Sponsor-Investigator, Qi Zhou, Academic leaders of Gynecologic Oncology Department, Chongqing University Cancer Hospital
Organization: Chongqing University Cancer Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CQGOG0401
Record Dates: First submitted 2021-08-04; First posted 2021-08-10 (Actual); Last update posted 2021-08-10 (Actual); Status verified 2021-08

CONDITIONS: 1. Relapsed Ovarian Cancer 2. Metastatic Ovarian Cancer 3. Endometrial Cancer 4. Cervical Cancer
MeSH Terms: conditions — Ovarian Neoplasms; Endometrial Neoplasms; Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ATG-008 + Chemotherapeutics (Experimental): ATG-008: Oral, 30 mg QD+Paclitaxel: 175 mg/m2, intravenous infusion >3 h, Day 1, Q3W; ATG-008: Oral, 30 mg QD+Carboplatin: AUC = 5, intravenous infusion >1 h, Day 1, Q3W or Cisplatin: 75 mg/m2, intravenous infusion >1h, Day 2, Q3W ; ATG-008: Oral, 30 mg QD+Doxorubicin hydrochloride liposome, 40 mg/m2, Day 1; Q4W;
  Interventions: Drug: ATG-008
- ATG-010 + Chemotherapeutics (Experimental): perimental: ATG-010 + Chemotherapeutics ATG-010: Oral, 80 mg QW, Day 1/week of treatment cycles +Paclitaxel: 175 mg/m2, intravenous infusion >3 h, Day 1, Q3W; ATG-010: Oral, 80 mg QW, Day
  1/week of treatment cycles +Carboplatin: AUC = 5, intravenous infusion >1 h, Day 1, Q3W or Cisplatin: 75 mg/m2, intravenous infusion >1h, Day 2, Q3W ; ATG-010: Oral, 80 mg QW, Day 1/week of treatment cycles +Doxorubicin hydrochloride liposome, 40 mg/ m2, Day 1; Q4W;
  Interventions: Drug: ATG-010

INTERVENTIONS:
Drug: ATG-008 — ATG-008 will be orally administered at 30 mg QD combined with chemotherapies. And about 8-12 subjects plan in each cohort.
  Arms: ATG-008 + Chemotherapeutics
Drug: ATG-010 — ATG-010 will be orally administered at 30 mg QD and 80 mg QW combined with chemotherapies. And about 8-12 subjects plan in each cohort.
  Arms: ATG-010 + Chemotherapeutics

SUMMARY:
1. This is a multi-center clinical study to evaluate dual mTORC1/2 inhibitor (ATG 008) or selective inhibitor of nuclear export compound (ATG-010) in combination with chemotherapy in patients with relapsed or metastatic ovarian cancer, endometrial cancer, and cervical cancer.

DETAILED DESCRIPTION:
This is a multi-center clinical study to evaluate dual mTORC1/2 inhibitor (ATG 008) or selective inhibitor of nuclear export compound (ATG-010) in combination with chemotherapy in patients with relapsed or metastatic ovarian cancer, endometrial cancer, and cervical cancer. And two cohorts of ATG-008 30 mg QD or ATG-010 80 mg QW in combination with chemotherapy will enroll subjects with platinum-sensitive ovarian cancer, platinum-resistant ovarian cancer, endometrial cancer, and cervical cancer, with about 8-12 subjects in either cohort. A total of about 64-96 subjects plan to be enrolled.

ELIGIBILITY:
Inclusion Criteria:

1. Understand and voluntarily sign informed consent (ICF).
2. Age 18 to 70 (including 18 and 70).
3. Histopathological or clinical diagnosis of high grade relapsed or metastatic serous ovarian cancer (including fallopian tube cancer and peritoneal cancer), endometrial cancer (including endometrial carcinosarcoma) and cervical cancer (squamous cell carcinoma, adenocarcinoma, and adenosquamous carcinoma); received ≤1 line treatment after recurrence.
4. At least one measurable lesion as defined by Response Evaluation Criteria in Solid Tumors (RECIST) v1.1.
5. Eastern Cooperative Oncology Group (ECOG) performance status 0 or

1. 6. Life expectancy >3 months. 7. Women of childbearing potential must agree to use effective contraceptives from signing the informed consent until 180 days after the last dose of study drug. Women of childbearing age include premenopausal women and women within 2 years after menopause. Women of childbearing age must have a negative blood pregnancy test at screening

Exclusion Criteria:

* 1. Histopathological diagnosis of sarcoma, carcinosarcoma (except endometrial carcinosarcoma). 2. Low-grade serous carcinoma, clear cell carcinoma, and mucinous carcinoma. 3. Symptomatic central nervous system metastases (except those who have been previously treated for brain metastases but have been keeping stable of disease status for 4 weeks prior to screening). 4. Participated in other clinical trials within 4 weeks prior to screening. 5. Received major surgery within 4 weeks prior to screening or expect to proceed a major surgical treatment during the study period. 6. Received systemic chemotherapy, radiotherapy, traditional Chinese medicine with anti tumor indications within 4 weeks prior to screening, or plan to receive therapeutic radiotherapy during the study period. 7. Received live attenuated vaccine within 4 weeks before screening, or plan to receive live attenuated vaccine during screening. 8. Using systemic immunosuppressive drugs currently or used within two weeks before screening with the following exceptions:

  1. Intranasal, inhaled, topical steroid or topical steroid injection (eg, intraarticular),
  2. Systemic corticosteroids at physiologic doses not to exceed 10 mg/ day of prednisone or equivalent, OR
  3. Steroids as premedication for hypersensitivity reactions (eg, computed tomography [CT] scan premedication). 9. Suffer from swallowing dysfunction, active gastrointestinal diseases or other diseases or disorders that affect the absorption, distribution, metabolism, and excretion of ATG-008 or ATG 010. 10. Hepatitis B virus (HBV) infection (Hepatitis B surface antigen [HBsAg] positive) or active hepatitis C virus (HCV) infection (HCVRNA positive at screening).

     11. Subjects with a history of human immunodeficiency virus (HIV) infection and/or acquired immunodeficiency syndrome. 12. Hypersensitive or known to be allergic to ATG-008, ATG-010 or chemotherapeutic agents or to active or inactive ingredients of drugs with similar chemical structures. 13. Have a history of organ transplantation (eg, liver transplantation or autologous stem cell transplantation). 14. Known as alcohol or drug dependent. 15. Female subjects who are pregnant or lactating. 16. Judgment by the investigator that the subject should not participate in the study by consideration of the complications or other conditions which might affect their adherence to the protocol.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2021-08-03 (Estimated); Primary Completion 2024-01-09 (Estimated); Study Completion 2024-04-09 (Estimated)

PRIMARY OUTCOMES:
Objective response rate(ORR) | 26 months
  Objective response rate(ORR)

SECONDARY OUTCOMES:
Time to response(TTR) | 26 months
  Evaluated by investigators according to RECIST 1.1
Duration of Response(DOR) | 26 months
  Evaluated by investigators according to RECIST 1.1
Disease control rate(DCR) | 26 months
  Evaluated by investigators according to RECIST 1.1
Overall Survival(OS) | 26 months
  The estimates of Kaplan-Meier
Progression-Free Survival(PFS) | 26 months
  Evaluated by investigators according to RECIST 1.1
The incidence,severity,and causality of AE,SAE | 26 months
  To evaluate the safety and tolerability of ATG-008 or ATG-010 in
EORTC-QLQ-C30 | 26 months
  To evaluate the safety and tolerability of ATG-008 or ATG-010 in

CONTACTS AND LOCATIONS:
Locations (1):
- Chongqing Cancer Hospital, Chongqing, Chongqing Municipality, China